CLINICAL TRIAL: NCT01669863
Title: Awake Extracorporeal Membrane Oxygenation (ECMO) for Acute Respiratory Failure A Non-controlled, Single-center, Investigator-initiated Prove-of-concept Study
Brief Title: Extracorporeal Membrane Oxygenation (ECMO) in Non-intubated Patients With Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Marius Hoeper, MD, Principle Investigator, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHH-6208
Record Dates: First submitted 2012-08-15; First posted 2012-08-21 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-03

CONDITIONS: ARDS
Keywords: ARDS
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of ECMO in non-intubated patients (Experimental): ECMO will be used in non-intubated patients with ARDS
  Interventions: Device: ECMO; Procedure: ECMO in non-intubated patients

INTERVENTIONS:
Device: ECMO — Use of veno-venous ECMO in non-intubated patients with ARDS
Procedure: ECMO in non-intubated patients — Use of veno-venous ECMO in non-intubated patients with ARDS

SUMMARY:
Proof-of-concept study addressing the feasibility of awake ECMO (v/v) in patients with acute respiratory failure

DETAILED DESCRIPTION:
Pilot study in 6 patients with ARDS addressing the use of awake veno-venous ECMO to avoid endotracheal intubation and mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 yrs with acute respiratory failure due to ARDS or pneumonia fulfilling standard criteria for endotracheal intubation

  * Severe and progressive hypoxemia, i.e. PaO2 < 60 mmHg or SaO2 < 90% on O2 > 10 l/min not tolerating noninvasive ventilation, or
  * PaO2/FiO2 < 200 not improving or deteriorating on noninvasive ventilation, or
  * Respiratory distress and hypoxemia not fulfilling the criteria above with clinical impression of the ICU attending that intubation and mechanical ventilation are mandated
* Patient considered eligible by at least two investigators of this study

Exclusion Criteria:

* Patient does not fulfill the inclusion criteria
* Uncontrolled malignancy
* Severe and untreatable coagulation or bleeding disorders (INR > 2,0; aPTT > 60s, Platelet count < 50.000/µl, all after substitution)
* Stroke within the past 3 months
* Uncontrolled sepsis or septic shock
* Multiorgan failure involving > 2 organ systems
* Norepinephrine dose > 1 mg/h
* Hyperdynamic circulation, indicated by cardiac index > 4.0 l/min/m2 (measured by PiCCO or Swan-Ganz catheter), or SvO2 > 80%
* Cardiac pump failure, indicated by echocardiography (EF < 40%), PiCCO or Swan Ganz catheter (CI < 2,5 l/min/m2 despite adequate volume management), or SvO2 < 50% (provided Hb > 9,0 g/dl and SaO2 > 90%), or the need for inotropes (dobutamine, epinephrine, levosimendan)
* Clinical or echocardiographic signs of pulmonary hypertension with right ventricular dysfunction
* APACHE-II score15 < 25
* Other conditions suggesting that the patient would benefit from intubation and mechanical ventilation
* Severe neurological disorders
* Estimated mortality due to severity of acute and/or underlying illness > 50%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius M Hoeper, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 patients recruited as planned
Groups:
- Use of ECMO in Non-intubated Patients: ECMO used in non-intubated patients with ARDS
  ECMO
  ECMO in non-intubated patients
Period: Overall Study
Arm/Group | Use of ECMO in Non-intubated Patients
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Use of ECMO in Non-intubated Patients: ECMO group
Arm/Group | Use of ECMO in Non-intubated Patients
Number analyzed (Participants) | 6
Age, Customized [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  Germany | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Did Not Require Endotrachael Intubation
Description: - N=6 patients will be enrolled in this exploratory pilot trial; if endotracheal intubation can be avoided in 2 or more of these patients, the trial will be considered positive. In that case, the next step would be a larger trial to better define the patient population with the highest likelihood of responding to this new therapeutic concept.
Time Frame: Duration of ICU stay
Measure: Number; unit: participants
Groups:
- Use of ECMO in Non-intubated Patients: ECMO will be used in non-intubated patients with ARDS
  ECMO
  ECMO in non-intubated patients
Arm/Group | Use of ECMO in Non-intubated Patients
Number analyzed (Participants) | 6
participants | 3

2. Secondary Outcome: Number of Participants Who Presented With ECMO-Related Complications
Description: ECMO-related complications
Time Frame: Duration of ICU stay
Measure: Number; unit: participants
Groups:
- Use of ECMO in Non-intubated Patients: ECMO in non-intubated patients
Arm/Group | Use of ECMO in Non-intubated Patients
Number analyzed (Participants) | 6
participants | 1

3. Other Pre Specified Outcome: Change in Oxygenation Index During Application of ECMO
Description: Oxygenation index (PaO2/FiO2) will be monitored regularly during the ICU stay
Time Frame: Duration of ICU stay
Population: Data for this outcome were not collected. We intended to measure the PaO2/FiO2 ratio in all patients anticipating that all patients would be mechanically ventilated, either invasively or non-invasively. However, it turned out that most patients did not require mechanical ventilation while on ECMO.
Arm/Group | Use of ECMO in Non-intubated Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Use of ECMO in Non-intubated Patients: Patients on ECMO
Arm/Group | Use of ECMO in Non-intubated Patients
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Use of ECMO in Non-intubated Patients (N=6)
Accidental ECMO line removal (Respiratory, thoracic and mediastinal disorders) | 1 — Patient intentionally removed his ECMO line

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes